CLINICAL TRIAL: NCT00008307
Title: Non-Ablative Chemotherapeutic Conditioning Before Allogeneic Stem Cell Transplantation
Brief Title: Combination Chemotherapy Followed by Donor Bone Marrow Transplant or Peripheral Stem Cell Transplant in Treating Patients With Hematologic Cancer or Genetic Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068396; CPMC-IRB-8462; CPMC-IRB-CAMP-25; NCI-G00-1897
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2006-04

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; chronic myelogenous leukemia, BCR-ABL1 positive; Philadelphia chromosome negative chronic myelogenous leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; intraocular lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; childhood chronic myelogenous leukemia; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Antilymphocyte Serum; Cyclosporine; fludarabine phosphate; Melphalan; Methylprednisolone; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Drug: methylprednisolone
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: syngeneic bone marrow transplantation

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as fludarabine and melphalan, before a donor bone marrow transplant or peripheral blood stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells and helps stop the growth of cancer or abnormal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy followed by donor bone marrow transplant or peripheral stem cell transplant works in treating patients with hematologic cancer or genetic disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the hematopoietic recovery in patients with hematologic malignancies or genetic disorders treated with fludarabine and melphalan followed by allogeneic or syngeneic bone marrow or peripheral blood stem cell transplantation.
* Determine the chemotherapeutic toxicity of this regimen in these patients.
* Determine the relapse and survival of patients treated with this regimen.
* Determine the incidence of graft-versus-host disease in patients treated with this regimen.

OUTLINE: Patients receive fludarabine IV on days -6 to -2 and melphalan IV on days -3 and -2. Patients with a non-HLA-identical family member may also receive anti-thymocyte globulin on days -4 to -1. Patients undergo allogeneic or syngeneic bone marrow or peripheral blood stem cell transplantation on day 0. Patients receive graft-vs-host disease prophylaxis comprising mycophenolate mofetil twice daily beginning on day -3, methylprednisolone beginning on day 5 and continuing over 8 weeks, and cyclosporine IV or orally beginning on day -3 and continuing until at least 6 months post-transplantation.

Patients are followed at 1, 3, and 6 months, and then at 1 year post-transplantation.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study within 5-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically and/or histologically confirmed hematologic malignancy or genetic disorder

  * Chronic myelogenous leukemia

    * Typical blood and marrow morphology
    * Presence of Philadelphia chromosome OR
    * Molecular evidence of bcr/abl rearrangement if Philadelphia chromosome-negative
  * Acute myeloid leukemia, acute lymphocytic leukemia, myelodysplasia, or lymphoma

    * High risk of relapse or progressive disease
    * Typical clinical features and morphology in blood, marrow, lymph node, or other tissue by cytochemistry, immunophenotyping, and/or chromosomal abnormalities
  * Multiple myeloma

    * Typical marrow morphology, radiographic findings, and paraprotein
  * Aplastic anemia

    * Typical marrow and blood findings
  * Genetic disorder including storage disease (e.g., adrenoleukodystrophy), hemoglobinopathies (e.g., thalassemia), or severe immunodeficiency
* Unwilling to undergo conventional high-dose chemoradiotherapeutic conditioning prior to allogeneic stem cell transplantation OR
* Presence of other medical disorder which precludes high-dose chemoradiotherapeutic conditioning (e.g., cardiac disease or infection)
* Syngeneic twin, HLA-identical, or 1 or 2 HLA antigen-mismatched family member or unrelated donor

PATIENT CHARACTERISTICS:

Age:

* 1 to 80

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other serious medical or psychiatric illness that would preclude study compliance
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 1998-04

PRIMARY OUTCOMES:
Hematopoietic recovery
Incidence of graft-versus-host disease

SECONDARY OUTCOMES:
Chemotherapeutic toxicity
Relapse and survival

CONTACTS AND LOCATIONS:
Overall Officials: David G. Savage, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States